CLINICAL TRIAL: NCT04331184
Title: Radiofrequency Ablation for Recurrent Hepatocellular Carcinoma After Locoregional Treatment Using Combined Bipolar and Monopolar Energy Deliver With Twin Cooled-Wet Electrodes: A Prospective Observational Study
Brief Title: RFA Using Combined Bipolar and Monopolar Energy Deliver With Twin Cooled-Wet Electrodes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-1907-157-1050
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Radiofrequency Ablation; Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RFA using combined bipolar and monopolar energy delivery (Experimental): Control group: The historic cohort is used to compare the results of the conventional alternating unipolar radiofrequency energy transfer mode with RFA.
  Interventions: Procedure: RFA using combined bipolar and monopolar energy deliver

INTERVENTIONS:
Procedure: RFA using combined bipolar and monopolar energy deliver — RFA technique combining bipolar mode and switching monopolar mode using dual / Twin Cooled-wet electrodes is performed on residual tumors after transarterial chemo-embolization.

SUMMARY:
In this study, a dual / Twin Cooled-wet electrode was used to perform RFA therapy on residual tumors after transarterial chemo-embolization and to find out the therapeutic results. The primary endpoint is the 12-month local recurrence rate, and the secondary endpoint is the survival rate, disease-free survival rate, actual procedure time, complications associated with the procedure, and the technical success rate for securing a safety margin of 3 mm or more around the tumor.

DETAILED DESCRIPTION:
In the treatment of HCC, local interventional procedures such as transarterial chemo-embolization and RFA are one of the most widely used methods. The probability of complete necrosis is known to be about 50-60% and 80%, respectively, and in a few cases, viable tumors remain, requiring additional treatment. Thus, in the treatment of residual tumors after locoregional intervention, RFA therapy is known as a safe and effective treatment, and in practice, it can be said to be a treatment that is often performed for the treatment of residual viable tumors. Until now, single or alternating monopolar mode and bipolar mode or multi-bipolar mode have been used for the transfer of radio frequency energy. Unipolar mode is used most frequnetly. Currently, in the present application, an alternating monopolar mode using three electrodes (Octopus electrode) and a bipolar mode using two electrodes (Twin cooled wet electrod, RF Medical) have been mainly used. RFA therapy for residual tumors after locoregional intervention has theoretically some limitations. First, it is difficult to deliver a sufficient amount of the high-frequency electrode per hour due to the high electrical resistance of the tissue due to tissue necrosis, fibrosis, and distribution of non-homogeneous tissue after local intervention. Second, the high frequency energy is distributed non-uniformly in the tissue. One of the ways to overcome this is to generate a high heat in the center and periphery of the tumor to be treated, a method of uniformly transmitting a large amount of energy such as high frequency or microwave, or a strategy to improve the thermal conductivity and electrical conductivity. In order to do this, saline is delivered to the high-frequency electrode to improve electrical conductivity, and at the same time, high-frequency energy can be applied to the center of the tumor and the periphery of the tumor if high-frequency energy can be transferred between the electrodes or around the two electrodes installed in the tumor. It can be evenly delivered and the efficiency of heat transfer is improved, which will improve the therapeutic effect of high-frequency heat therapy on residual tumors after local intervention.

Recently, Rf Medical in Korea has developed a twin cooled wet (TCW) electrode capable of injecting physiological saline into these high frequency electrodes and has been approved for clinical use under medical insurance. About 30% has been used using a bipolar mode, which has a theoretical advantage to concentrate high-frequency energy between the electrode and the electrode. However, according to the experience in the present application, when the bipolar mode is used, the rate of ablation is very fast and the transmission of high-frequency energy is relatively easy in the center of the tumor, but the transmission of high-frequency energy in the periphery of the tumor is relatively low, resulting in about 30% of tumors. A marginal recurrence or residual tumor was experienced in the margin, and in the last 6 months, bipolar mode and switching monopolar mode were combined to prevent recurrence in the periphery of the tumor, and treatment was performed with the default setting. The result is low recurrence (6 months local recurrence rate of about 15%).

ELIGIBILITY:
Inclusion Criteria:

* agree to the protocol's requirements and submit a consent form
* 20 years old-85 years old
* Child-Pugh Class A and B
* Patients with residual HCC after locoregional treatment who meet the following conditions A. Patients with a single nodular HCC within 5 cm or multiple nodular HCC of 3 or less in all cases of focal cancer B. Patients who did not have vascular invasion or extrahepatic metastasis during locoregional intervention

Exclusion Criteria:

* When the number of malignant HCC is 3 or more
* If the tumor has a maximum size of 3 cm or more
* diffuse infiltrative HCC
* Child-Pugh class C
* If there is an invasion of liver vessels due to malignant liver tumors
* severe coagulopathy
* multiple distant metastasis
* situations where it is very unlikely to obtain appropriate data for research purposes

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2020-01-28 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Local tumor progression | 12 months

SECONDARY OUTCOMES:
Overall survival rate | 12 months
  Survival data
Recurrence free survival | 12 months
  Survival data
Procedure time | immediately
  Procedure related outcome
complication rate | immediately
  Procedure related outcome
technical success rate | immediately
  Procedure related outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No